CLINICAL TRIAL: NCT04893525
Title: Evaluating Microdosing in Emergency Departments: A Randomized Controlled Trial Comparing the Effectiveness of Buprenorphine/Naloxone Microdosing vs. Standard Dosing (EMED Study)
Brief Title: Evaluating Buprenorphine/Naloxone Microdosing vs. Standard Dosing in Emergency Departments
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jessica Moe, Assistant Professor UBC Department of Emergency Medicine, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H20-03698
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Opioid-use Disorder
Keywords: Buprenorphine/naloxone; Suboxone; Opioid agonist treatment; Micro-induction; Microdosing
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive either a microdosing package or standard dosing package, using permuted blocks of variable sizes (2 and 4). We will stratify randomization by study site.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Buprenorphine/naloxone Microdosing (Active Comparator): Participants with Opioid use disorder will receive a Buprenorphine/naloxone microdosing package from the ED. This will consist of a five-day take-home packages with gradually increasing doses of 2mg/0.5mg buprenorphine/naloxone tablet employing a four times daily dosing schedule over five days.
  Day 1: Buprenorphine 0.5 mg-naloxone 0.125 mg SL* QID** (One quarter tablet),
  Day 2: Buprenorphine 1 mg-naloxone 0.25 mg SL QID (One half tablet),
  Day 3: Buprenorphine 2 mg-naloxone 0.5 mg SL QID (1 tablet),
  Day 4: Buprenorphine 3 mg-naloxone 0.75 mg SL QID (1.5 tablets)
  Day 5: Buprenorphine 16 mg-naloxone 4 mg SL once daily (8 tablets).
  *SL: Sublingual
  ** QID: four times daily
  Interventions: Drug: Buprenorphine/naloxone
- Buprenorphine/naloxone Standard Dosing (Active Comparator): The control intervention will be provision of a buprenorphine/naloxone standard dosing package from the ED. This will consist of a five day package with a commonly accepted standard dosing regimen aiming to achieve a therapeutic buprenorphine/naloxone dose within 24 hours of initiation. Standard dosing packages are currently available in EDs in BC and Alberta as standard of care.
  Day 1: Buprenorphine 2 mg-naloxone 0.5 mg SL q1h prn to a maximum of 6 tablets in the first 24 hours (1 tablet),
  Day 2: Buprenorphine 12 mg-naloxone 3 mg SL once daily (6 tablets),
  Day 3: Buprenorphine 16 mg-naloxone 3 mg SL once daily (8 tablets),
  Day 4:Buprenorphine 16 mg-naloxone 3 mg SL once daily (8 tablets).
  Day 5:Buprenorphine 16 mg-naloxone 3 mg SL once daily (8 tablets).
  Interventions: Drug: Buprenorphine/naloxone

INTERVENTIONS:
Drug: Buprenorphine/naloxone — Buprenorphine/naloxone is a first line, evidence-based opioid agonist therapy that improves mortality for people with opioid use disorder, and that has been demonstrated to be effective at retaining people in addictions care and decreasing illicit opioid use when initiated from EDs.
  Other Names: Suboxone

SUMMARY:
This is a multi-centre, open-label RCT at four Emergency Departments (EDs) in British Columbia and Alberta. The purpose of the current study is to compare the effectiveness of buprenorphine/naloxone microdosing and standard dosing take-home induction regimens at enabling patients to successfully complete the induction regimen, and at retaining patients on opioid agonist therapy.

We will randomize our enrolled patients to receive take-home microdosing or standard dosing packages of buprenorphine/naloxone. For the microdosing arm, patients immediately start taking low doses that increase to effective levels without requiring them to go into withdrawal.

We hypothesize that ED patients provided buprenorphine/naloxone microdosing packages will be more likely to successfully complete the induction period compare to patients provided standard dosing packages. We furthermore hypothesize that those provided microdosing will be more likely to be retained in opioid agonist therapy, and will experience lower overdose, mortality, and healthcare utilization subsequent to their ED visit.

DETAILED DESCRIPTION:
This multi-centered, open-label RCT will be carried out at four emergency departments (EDs) across Canada, two in British Columbia (Vancouver General Hospital and St. Paul's Hospital) and two in Alberta (Royal Alexandra Hospital and Northeast Health Centre). The investigators will randomize the selected patients to receive take-home microdosing or standard dosing packages. These will include a five-day regimen in a bubble package, along with over-the-counter adjunctive medication. The details of the different regimens are outlined in the "Study Arms" section of this page, and the adjunctive medication regimen is highlighted below.

The primary objective of the current study is to compare the effectiveness of ED-initiated buprenorphine/naloxone take-home standard dosing and microdosing interventions for patients with opioid use disorder identified at the four study ED's, with regard to a) successful completion of the induction period (primary outcome) and b) retention on opioid agonist therapy at 30, 90, and 365 days following ED visit, or decreasing overdose, mortality and healthcare utilization (secondary outcomes).

The primary outcome measure will be whether the patient filled a prescription for buprenorphine/naloxone within two weeks of their ED visit (binary variable). If this occurs, the investigators presume that the patient successfully completed the induction regimen provided, followed up with a healthcare provider able to prescribe buprenorphine/naloxone, and was subsequently prescribed ongoing buprenorphine/naloxone therapy. The investigators chose a two-week period, recognizing that patients receiving take-home packages from the ED may not start taking the induction regimen immediately after the ED visit, but instead may decide to delay the start of their regimen to a time that is more convenient to them. The investigators hypothesize that most patients would decide to start within two weeks of their ED visit. This hypothesis is supported by peer advisors on the study team.

Secondary outcomes will include retention on OAT, which will be assessed using provincial pharmacy records (PharmaNet and PIN) up to 30, 90 and 365 days.

The investigators will also examine fatal or non-fatal overdose, mortality, ED visits, physician visits, admissions, and days admitted within 30, 90 and 365 days (timeframes plausibly attributable to ED interventions). The investigators expect that successful OAT initiation would lead to decreased healthcare use, consistent with our previous work indicating high admissions among persons with recent OUD diagnoses and OAT discontinuation. The investigators will also assess patients' self-reported experiences with study regimens, withdrawal, precipitated withdrawal, and comfort via participant surveys.

The study will offer co-interventions to both the intervention and control groups that will be outlined in study-related pre-printed clinical ordersets. This will include symptomatic treatment of nausea/vomiting (dimenhydrinate: 50 mg PO q6h prn - 6 doses), and pain or myalgias (acetaminophen: 975 mg po q6h prn - 6 doses) (ibuprofen: 400 mg po q6h prn - 6 doses), to use in the first two days of inductions, when the investigators expect withdrawal symptoms to be most challenging, especially for standard dosing. Those receiving microdosing may experience breakthrough withdrawal if they do not take an adequate dose of overlapping opioid. Of note, enrolled patients will also be offered counselling with ED social workers to aid with social or other patient needs (e.g., housing, transportation).

This RCT builds on interventions, recruitment, and follow-up procedures successfully tested in a feasibility study. The study team has expertise in emergency and addictions medicine, peer engagement, community overdose prevention, biostatistics, health economics, and RCT implementation, including the high-profile SALOME trial comparing heroin and hydromorphone treatments in our target population. Knowledge users from provincial health ministry and regions will ensure scale-up. The study team are engaging people with lived experience throughout study design, implementation, and interpretation to ensure relevance.

The investigators will ascertain our primary and secondary outcome measures relating to completion of induction and retention on OAT, on records of prescriptions filled in provincial pharmacy databases: PharmaNet in BC, and the Pharmaceutical Information Network in Alberta. The investigators specifically selected partner sites in BC and Alberta to allow our team to access these provincial administrative databases for outcome ascertainment, which will minimize losses to follow-up and strengthen the reliability of our results. The investigators will assess secondary outcomes of overdose and mortality by linking our study cohort to the BC Centre for Disease Control Overdose Cohort (for patients enrolled in BC), and to provincial Vital Statistics data (Alberta and BC). The investigators will assess secondary outcomes related to healthcare utilization by linking our study cohort to provincial databases on emergency department visits (National Ambulatory Care Reporting System) and hospitalizations (Discharge Abstract Data) in Alberta and BC. We will access all administrative databases through Population Data BC (PopData BC) and Alberta Health Services.

This trial will inform urgent development of effective ED buprenorphine/naloxone programs to improve OAT access for people at high risk of overdose. The investigators will leverage our networks of policy makers, public health leaders, and health providers to enable rapid dissemination of findings in guidelines and policies across Canada.

ELIGIBILITY:
Inclusion Criteria:

We will include ED patients ≥18 years of age with opioid use disorder who are being discharged from the ED. We will define opioid use disorder as non-medical opioid use in the previous 30 days and a positive score for opioid dependency based on the validated Rapid Opioid Dependence Screen (RODS).

All patients will also be assessed by the treating physician or degree of clinical opioid withdrawal, based on the clinical opiate withdrawal scale (COWS) score. Patients will be eligible for the take-home study interventions if they have a COWS score <=12, as a score greater than 12 would mean the patient is a candidate for standard buprenorphine induction in the ED at that moment in time, and would therefore not be eligible for outpatient study interventions.

Exclusion Criteria:

* Active withdrawal at time of ED assessment (Clinical Opiate Withdrawal Score [COWS] >12)
* Admitted to hospital
* Severe communication barriers that inhibit patients' understanding of study procedures and interventions
* Are taking opioids for cancer or palliative-care related indications
* Are deemed unsafe to approach by ED providers
* Incarceration
* Not a resident of the province in which they are seeking care (BC or Alberta)
* Actively receiving OAT, defined as having filled a prescription for one of the following medications in the 5 days prior to ED presentation: buprenorphine/naloxone, methadone, sustained release morphine, injectable hydromorphone, injectable diacetylmorphine
* Prior enrollment in the study
* Known or suspected mechanical gastrointestinal obstruction (e.g., bowel obstruction or strictures) or any diseases/conditions that affect bowel transit (e.g., ileus of any type).
* Suspected surgical abdomen (e.g., acute appendicitis or pancreatitis).
* Severe respiratory insufficiency.
* Severe CNS depression, increased cerebrospinal or intracranial pressure, and head injury.
* Complicating patient factors that make home inductions from the ED unsafe and/or that require expert consultation for consideration of induction in an observed setting.

These factors include:

* Allergy to buprenorphine/naloxone
* Severe respiratory or liver dysfunction
* Concurrent withdrawal or intoxication from sedatives (e.g., alcohol, benzodiazepines)
* Active prescription for sedative medications (e.g., benzodiazepines, opioids)
* Use of monoamine oxidase inhibitors within the past 14 days
* Concerns that the patient is unable to safely store medications
* Pregnancy (we will obtain a point-of-care urine pregnancy test on all women of child-bearing age prior to enrollment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 658 (Estimated)
Dates: Start 2021-07-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients who have filled a prescription for buprenorphine/naloxone within two weeks of their ED visit. | 14 days
  Number of patients who have filled a prescription for buprenorphine/naloxone within two weeks of their ED visit.

SECONDARY OUTCOMES:
Number of patients retained in Opioid agonist therapy (OAT) following the ED visit | 30, 90, and 365 days
  Number of patients retained in Opioid agonist therapy (OAT) following the ED visit
Number of fatal or non-fatal overdose events, mortality, ED visits, physician visits, admissions, and days admitted to hospital for patients following ED visit. | 30, 90, and 365 days.
  Number of fatal or non-fatal overdose events, mortality, ED visits, physician visits, admissions, and days admitted to hospital for patients following ED visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Moe, MD, Principal Investigator — University of British Columbia
Locations (6):
- Canada (6):
  - Foothills Medical Centre, Calgary, Alberta
  - Northeast Community Health Centre, Edmonton, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - University of British Columbia Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers

REFERENCES:
- [Background] Moe J, Badke K, Pratt M, Cho RY, Azar P, Flemming H, Sutherland KA, Harvey B, Gurney L, Lockington J, Brasher P, Gill S, Garrod E, Bath M, Kestler A. Microdosing and standard-dosing take-home buprenorphine from the emergency department: A feasibility study. J Am Coll Emerg Physicians Open. 2020 Oct 20;1(6):1712-1722. doi: 10.1002/emp2.12289. eCollection 2020 Dec. PMID 33392580
- [Background] Moe J, Doyle-Waters MM, O'Sullivan F, Hohl CM, Azar P. Effectiveness of micro-induction approaches to buprenorphine initiation: A systematic review protocol. Addict Behav. 2020 Dec;111:106551. doi: 10.1016/j.addbeh.2020.106551. Epub 2020 Jul 11. PMID 32739588
- [Background] Moe J, O'Sullivan F, Hohl CM, Doyle-Waters MM, Ronsley C, Cho R, Liu Q, Azar P. Short communication: Systematic review on effectiveness of micro-induction approaches to buprenorphine initiation. Addict Behav. 2021 Mar;114:106740. doi: 10.1016/j.addbeh.2020.106740. Epub 2020 Nov 25. PMID 33352498